CLINICAL TRIAL: NCT06233838
Title: Prospective, Multicenter, Randomized, Open Label Study on the Efficacy and Safety of Comparison of KHA80 Blood Perfusion Combined With Hemodialysis and Conventional Hemodialysis in Clearing IL-6, β2-MG and PTH in Maintenance Hemodialysis Patients
Brief Title: Multi-center Clinical Study on Hemoperfusion of KHA80
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, wanjianxin, Clinical Professor, First Affiliated Hospital of Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8339-001
Record Dates: First submitted 2024-01-08; First posted 2024-01-31 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Uremia; Uremic Osteodystrophy; Dialysis Related Complication
Keywords: KHA80; Maintenance hemodialysis; IL-6; β2-MG; PTH
MeSH Terms: conditions — Uremia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KHA80 hemoperfusion treatment (Experimental): The experimental group (197 cases) were randomly assigned to receive Jianfan KHA80 hemoperfusion treatment on the basis of hemodialysis or hemodiafiltration treatment, and the frequency of hemoperfusion treatment was ≥2 times/month.
  Interventions: Device: KHA80 hemoperfusion treatment
- Routine hemodialysis (No Intervention): Randomly assign the control group (197 cases) to receive hemodialysis or hemodialysis filtration treatment, and the frequency of treatment is ≥2 times/week.

INTERVENTIONS:
Device: KHA80 hemoperfusion treatment — On the basis of hemodialysis or hemodiafiltration treatment, Jianfan KHA80 hemoperfusion treatment was given, and the frequency of hemoperfusion treatment was ≥2 times/month.
  Arms: KHA80 hemoperfusion treatment

SUMMARY:
To evaluate the decreasing rate of blood IL-6, β2-MG and PTH in maintenance hemodialysis patients in the 52nd week compared with routine hemodialysis.

DETAILED DESCRIPTION:
394 patients with maintenance hemodialysis were included in the study, and the blood purification time was ≥8 hours per week (including routine hemodialysis, high-throughput hemodialysis, hemodialysis filtration, hemoperfusion, etc.). Randomly assign the control group (197 cases) to receive hemodialysis or hemodialysis filtration treatment, and the frequency of treatment is ≥2 times/week; The experimental group (197 cases) were randomly assigned to receive Jianfan KHA80 hemoperfusion treatment on the basis of hemodialysis or hemodiafiltration treatment, and the frequency of hemoperfusion treatment was ≥2 times/month. The follow-up data of 0, 4, 12, 24, 36 and 52 weeks of treatment in the two groups were collected, and the information of combined medication and adverse events was also collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, regardless of sex;
2. According to the 2012 KDIGO guidelines, it was diagnosed as CKD5 (EGFR ≦ 15ml/(min ˙ 1.73m2));
3. receive regular hemodialysis (including hemodialysis filtration) for 4 hours twice a week for ≧3 months;
4. blood β 2-mg ≥ 30 mg/L and/or PTH ≥ 600 pg/mL and/or IL-6 ≥ 16.2 pg/mL;
5. Sign the informed consent form.

Exclusion Criteria:

1. Those who are known to have allergic reactions, contraindications or intolerance to the materials of dialyzers and hemoperfutors;
2. Patients with severe bleeding tendency and active bleeding, or with definite coagulation dysfunction, with a platelet count of < 60× 109/L;
3. Hemodialysis blood flow < 200 ml/min.
4. Kt/V<1.2；
5. Serum albumin < 30g/L;
6. Parathyroid resection within one year;
7. people with low blood pressure and severe cardiopulmonary insufficiency;
8. lactating or pregnant women or those who plan to be pregnant within one year;
9. infection, history of malignant tumor, active stage of rheumatic immune disease;
10. Patients whose life expectancy is less than one year;
11. Other clinical researchers are currently or recently (within 30 days);
12. According to the researcher's judgment, the patient has other unsuitable conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2025-01-13 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
the rate of change of IL-6, β2-MG and PTH | in the 52nd week
  the rate of change of IL-6, β2-MG and PTH in the 52nd week of maintenance hemodialysis patients compared with routine hemodialysis.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen SJ, Jiang GR, Shan JP, Lu W, Huang HD, Ji G, Wu P, Wu GF, Wang W, Zhu C, Bian F. Combination of maintenance hemodialysis with hemoperfusion: a safe and effective model of artificial kidney. Int J Artif Organs. 2011 Apr;34(4):339-47. doi: 10.5301/IJAO.2011.7748. PMID 21534244
- [Background] Kaysen GA. The microinflammatory state in uremia: causes and potential consequences. J Am Soc Nephrol. 2001 Jul;12(7):1549-1557. doi: 10.1681/ASN.V1271549. PMID 11423586
- [Background] Rao M, Guo D, Perianayagam MC, Tighiouart H, Jaber BL, Pereira BJ, Balakrishnan VS. Plasma interleukin-6 predicts cardiovascular mortality in hemodialysis patients. Am J Kidney Dis. 2005 Feb;45(2):324-33. doi: 10.1053/j.ajkd.2004.09.018. PMID 15685511
- [Background] Thang LV, Loc ND, Dung NH, Kien NT, Quyen DBQ, Tuan NM, Ha DM, Kien TQ, Dung NTT, Van DT, Van Duc N, Ha NTT, Toan PQ, Usui T, Nangaku M. Predicting 3-year mortality based on the tumor necrosis factor alpha concentration in low-flux hemodialysis patients. Ther Apher Dial. 2020 Oct;24(5):554-560. doi: 10.1111/1744-9987.13463. Epub 2020 Jan 27. PMID 31856402
- See also: Combination of maintenance hemodialysis with hemoperfusion: a safe and effective model of artificial kidney — http://pubmed.ncbi.nlm.nih.gov/21534244/
- See also: The microinflammatory state in uremia: causes and potential consequences. — http://pubmed.ncbi.nlm.nih.gov/11423586/
- See also: Plasma interleukin-6 predicts cardiovascular mortality in hemodialysis patients — http://pubmed.ncbi.nlm.nih.gov/15685511/
- See also: Predicting 3-year mortality based on the tumor necrosis factor alpha concentration in low-flux hemodialysis patients — http://pubmed.ncbi.nlm.nih.gov/31856402/

DOCUMENTS (1):
  • Informed Consent Form (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT06233838/ICF_000.pdf